CLINICAL TRIAL: NCT04263077
Title: The Effect of Kinesio Taping Tension on the Pressure-pain Threshold and Pain Tolerance: a Randomized Controlled Trial
Brief Title: The Effect of Kinesio Taping Tension on the Pain Threshold and Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, OYKU AVCI, GRADUATE STUDENT, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 180176
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: PRESSURE PAIN THRESHOLD; PAIN TOLERANCE; KINESIOTAPING
Keywords: KINESIOTAPING

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PLACEBO (Placebo Comparator): IN THE PLACEBO GROUP, THE ENDS OF THE TAPES WILL BE APPLIED NO TENSION WITHOUT OVERLAPPING EACH OTHER.
  Interventions: Other: PLACEBO
- 50% TENSION GROUP (Other): KINESIOTAPE WILL BE APPLIED WITH 50% TENSION.
  Interventions: Other: 50% TENSION GROUP
- 75% TENSION GROUP (Other): KINESIOTAPE WILL BE APPLIED WITH 75% TENSION.
  Interventions: Other: 75% TENSION GROUP
- 100% TENSION GROUP (Other): KINESIOTAPE WILL BE APPLIED WITH 100% TENSION.
  Interventions: Other: 100% TENSION GROUP

INTERVENTIONS:
Other: PLACEBO — The diamond shape technique, which is a kinesio tape technique, will be used in the lateral epicondyle region. The ends of the kinesiotapes will be applied tension-free without overlapping.
  Arms: PLACEBO
Other: 50% TENSION GROUP — Kinesiotape will be applied to the lateral epicondyle region with 50% tension.
  Arms: 50% TENSION GROUP
Other: 75% TENSION GROUP — Kinesiotape will be applied to the lateral epicondyle region with 75% tension.
  Arms: 75% TENSION GROUP
Other: 100% TENSION GROUP — Kinesiotape will be applied to the lateral epicondyle region with 100% tension.
  Arms: 100% TENSION GROUP

SUMMARY:
The aim of this study was to investigate the effects of kinesiotape technique applied in different tensions on pain tolerance (PT) of healthy university students. 100 healthy and volunteer male individuals studying at Mugla Sitki Kocman University Faculty of Health Sciences will participate in the research. Study protocol was approved by the ethics committee of Mugla Sitki Kocman University. The study is designed as a randomized, controlled, double-blind study to be performed on 4 groups consisting of 25 individuals in each group (No tension(Placebo), and 50%, 75%, 100% tensions of Kinesiotape). Kinesiotape will be applied over lateral epicondyle of the dominant extremities with diamond shape technique by a KTAI®certified physiotherapist. PT's will be measured with J-Tech algometer before, immediately and 30 minutes after taping by a different physiotherapist who will be blind to taping tension.

DETAILED DESCRIPTION:
Diamond shape banding method will be applied in a way that 4 bands of 2.5 cm width cut kinesio tape ends on top of each other, leaving the lateral epicondyle region exposed while the elbows are slightly flexed in the supine position. In the groups where different tensions will be applied, the middle points of the tapes will be stretched according to the amount of tensions, and the ends will be taped over each other without tension.In the placebo group, the tapes of the tapes will be applied tensionlessly without overlapping each other. Algometer will be used in the assessment of pressure pain threshold and pain tolerance. Pain severity felt at the level of pain threshold and pain tolerance will be evaluated with the Visual Analogue Scale (VAS). All measurements will be made before taping, immediately after taping and 30 minutes after taping, will be repeated 3 times and their average values will be recorded. There will be a 60 second rest period between each trial to avoid temporal sensitization. Each assessment will be performed bilaterally by another physiotherapist who is blind to the band tension and has no experience with the kinesio banding technique.

ELIGIBILITY:
Inclusion Criteria:

* Being a male university student over the age of 18
* Volunteering for the study
* Filling out the informed consent form Not having the knowledge and experience about kinesiotaping before

Exclusion Criteria:

* Being diagnosed with lateral epicondylit and its treatment
* Having any neurological disease or systemic disease that disrupts sense / pain perception (diabetes, rheumatoid arthritis, peripheral vascular disease, etc.)
* Skin sensitivity to elastic banding
* Open wound, ulcer, fungal infection in the area to be taped
* Exposure to upper extremity and / or cervical injury in the past 6 months

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | 10 minutes
  Study will be performed with 4 groups of 25 individuals, each of whom use the kinesiotape at different tensions. 0% tension application will be for Placebo, 50% tension application, 75% tension application 100% tension application. In groups with different tension banding, pressure pain threshold will be measured with algometer bilaterally. Measurements will be repeated 3 times and their average will be recorded.
Pain Tolerance | 10 minutes
  After measuring the pressure pain threshold, the pain tolerance of the same groups will be measured with an algometer. Measurements will be repeated 3 times and their average will be recorded.
Visual Analog Scale | 10 minutes
  Pain severity felt at the level of pain threshold and pain tolerance will be evaluated with the Visual Analogue Scale (VAS) bilaterally. The pain intensity created by the algometer probe end will be measured by VAS. The patients will mark the severity of their pain on a 100 mm line, one end of which is painless and the other end expressing unbearably severe pain. Values close to 0 mean that the pain is less, and values close to 100 indicate that the pain is high.The VAS assessment will be done immediately after each pressure pain threshold and pain tolerance measurements. Measurements will be repeated 3 times and their average will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Tuğay, PhD, Study Chair — Muğla Sıtkı Koçman University
Locations (1):
- Mugla Sitki Kocman University Health Sciences Faculty, Muğla, Turkey (Türkiye)